CLINICAL TRIAL: NCT01297907
Title: Bronchial Hyperreactivity in Children With Crohn Disease
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof. Lea Bentur, Rambam Health Care Campus
Other Study IDs: Crohn's
Record Dates: First submitted 2011-01-24; First posted 2011-02-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2007-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Bronchial hyper reactivity; Fractional exhaled NO; Methacholine Challenge Test; Pediatric Crohn's Disease Activity Index; To determine the frequency of bronchial hyperreactivity in pediatric patients followed and treated for Crohn disease
MeSH Terms: conditions — Crohn Disease | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Crohn's Patients: Random Crohn's Disease Patients that can perform Methacholine Challenge Test (MCT)
  Interventions: Other: Methacholine Challenge Test; Other: Fractional Exhaled NO (FENO); Other: Blood Test; Other: PCDAI
- Negative MCT: Patients evaluated for functional cough who had negative Methacholine Challenge Test (MCT)
  Interventions: Other: Methacholine Challenge Test; Other: Fractional Exhaled NO (FENO)

INTERVENTIONS:
Other: Methacholine Challenge Test — Methacholine challenge test to evaluate airway hyperreactivity
Other: Fractional Exhaled NO (FENO) — Fractional Exhaled NO to evaluate eosinophilic inflammation
Other: Blood Test — Blood Tests (Eosinophil Count)
  Groups: Crohn's Patients
Other: PCDAI — Clinical Evaluation for Pediatric Crohn's Disease Activity Index (PCDAI)
  Groups: Crohn's Patients

SUMMARY:
Background: Latent pulmonary involvement is described in Crohn Disease(CD). Bronchial hyperreactivity measured by the Methacholine Challenge Test (MCT) has been evaluated in two studies involving mainly adults.Our aim was to determine the frequency of bronchial hyperreactivity in pediatric patients followed and treated for Crohn disease.

Methods: Twenty-three children with Crohn disease completed a questionnaire, followed by spirometry, Methacholine Challenge Test (MCT) and determination of Fractional Exhaled NO (FENO). The control group included patients evaluated for functional cough who had negative Methacholine Challenge Test (MCT).

ELIGIBILITY:
Inclusion Criteria:

* Children with Crohn disease
* Children that can perform lung function tests (MCT)

Exclusion Criteria:

* Upper respiratory tract infection last month
* Fever or Pneumonia last month
* Smoking
* Other chronic diseases
* Other respiratory diseases

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Twenty-three children with Crohn disease in the age of 11 to 22 yr
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Methacholine challenge test | 18 months
  As assessed by methacholine challenge test with determination of PC20.

SECONDARY OUTCOMES:
Fractional Exhaled NO | Day 1
  Exhaled NO test
Eosinophils count | Day 1
  blood test
Pediatric Crohn's Disease Activity Index (PCDAI) | Day 1
  Clinical Evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel